CLINICAL TRIAL: NCT04675918
Title: Pediatric In-Hospital Cardiac Arrest International Registry (PACHIN): a Prospective International Multicenter Register of Cardiac Arrest in Children.
Brief Title: Pediatric In-Hospital Cardiac Arrest International Registry (PACHIN)
Acronym: PACHIN
Status: Recruiting | Type: Observational
Sponsor: Jimena del Castillo (Other)
Responsible Party: Sponsor-Investigator, Jimena del Castillo, MD, PhD, Hospital General Universitario Gregorio Marañon
Organization: Hospital General Universitario Gregorio Marañon (Other)
Other Study IDs: ESCE-RCP 2.0; PI18/01632 (Other Grant/Funding Number: ISCIII)
Record Dates: First submitted 2020-11-27; First posted 2020-12-19 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Cardiac Arrest; Pediatric ALL; In-hospital Cardiac Arrest
Keywords: pediatric cardiac arrest; outcomes; survival; cardiopulmonary resuscitation
MeSH Terms: conditions — Heart Arrest; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Heart Arrest, Induced

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Cardiac arrest — Definition of characteristics of cardiac arrest and resuscitation as well as post-resuscitational care and follow up.

SUMMARY:
: An intrahospital CA data recording protocol has been designed following the Utstein model. Database is hosted according to European legislation regarding patient data protection. It is drafted in English and Spanish. Invitation to participate has been sent to Spanish, European and Latinamerican hospitals. Variables included, asses hospital characteristics, the resuscitation team, patient's demographics and background, CPR, post-resuscitation care, mortality, survival and long-term evolution. Survival at hospital discharge will be evaluated as a primary outcome and survival with good neurological status as a secondary outcome, analyzing the different factors involved in them

DETAILED DESCRIPTION:
Study design: this study is a multicenter, international, prospective observational registry.

Setting: patients will be enrolled by participating investigators from European and Latinamerican countries. All sites are susceptible of treating pediatric cardiac arrest patients. Participating hospitals differ in levels of care but are all able to submit their data to the study's database.

Patient elegibility: Inclusion criteria: all children aged 1 month to 18 years who suffer a CA in hospital. For the study, CA is defined as the absence of vital signs requiring at least one minute of chest compressions. Subsequent episodes of CA may be included for the same individual.

Exclusion criteria: Patients being treated with extracorporeal circulatory support (ECMO or ventricular assistance) at the time of CA. Patients who suffer a cardiac arrest and require ECMO for ROSC, after performing conventional CPR, will not be excluded. Duration of the data collection period 24 months.

Recruitment: Study candidates will be identified by a study physician, who will explain the study to parents or guardians. Written informed consent will be obtained from parents or guardians prior to inclusion in the study. A CONSORT (Consolidated Standard of Reporting Trials) flow diagram is shown in Figure 1.

Data collection: data will be collected, verified, and uploaded to a protected electronic web-based database (Xolomon) by their designated site coordinators/investigators under the oversight of their IRB. Database has been designed following the Utstein model (19). Database is hosted according to European legislation regarding patient data protection. It is drafted in English and Spanish.

ELIGIBILITY:
Inclusion Criteria:

* all children aged 1 month to 18 years who suffer a CA in hospital

Exclusion Criteria:

* Patients being treated with extracorporeal circulatory support (ECMO or ventricular assistance) at the time of CA.
* Duration of resuscitation < 1minute

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patients who suffer a cardiac arrest in hospital premises and are resuscitated with at least 1 minute of cardiopulmonary resuscitation measures.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Survival | Through study completition an average of 3 years
  Survival

SECONDARY OUTCOMES:
Neurological outcome | 5 years
  Neurological outcome (Scales: Pediatric Cerecral Performance Category Scale and Pediatric Overall Performance Category Scale. Assesment of neurological outcome with both scales which attempt to measure the same items in neurological development in pediatric patients. Values of 1 or 2 describe normal recovery whilst values of 5-6 define brain death.

CONTACTS AND LOCATIONS:
Locations (1):
- Gregorio Marañon Hospital, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Del Castillo J, Sanz D, Herrera L, Lopez-Herce J; Grupo de Estudio de Parada Cardiaca Intrahospitalaria en la Infancia. Pediatric In-Hospital Cardiac Arrest International Registry (PACHIN): protocol for a prospective international multicenter register of cardiac arrest in children. BMC Cardiovasc Disord. 2021 Jul 31;21(1):365. doi: 10.1186/s12872-021-02173-5. PMID 34332522